CLINICAL TRIAL: NCT06155773
Title: Effect of Cervical Margin Relocation With Different Restorative Materials on Three-year Clinical Performance and In-Vitro Fracture Resistance of Indirect Hybrid Ceramic Onlay Restorations
Brief Title: Clinical Performance of Onlay Restorations After Cervical Margin Relocation (CMR)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Mansoura University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 9153193
Record Dates: First submitted 2023-10-17; First posted 2023-12-04 (Actual); Last update posted 2023-12-08 (Actual); Status verified 2023-05

CONDITIONS: Dental Caries
MeSH Terms: conditions — Dental Caries

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: double blind
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Highly viscous Glass Ionomer (Experimental): Highly viscous glass ionomer restoration is used to elevate the subgingival cervical margin in deep class II cavities before receiving cad/cam onlay restoration
  Interventions: Procedure: Highly viscous glass ionomer (cervical margin relocation)
- Low shrinkage Flowable Composite (Experimental): Low shrinkage Flowable Composite restoration is used to elevate the subgingival cervical margin in deep class II cavities before receiving cad/cam onlay restoration
  Interventions: Procedure: Low shrinkage Flowable Composite (cervical margin relocation)
- Resin Modified Glass Ionomer (Experimental): Resin Modified Glass Ionomer restoration is used to elevate the subgingival cervical margin in deep class II cavities before receiving cad/cam onlay restoration
  Interventions: Procedure: Resin Modified Glass Ionomer (cervical margin relocation)
- Bioactive Ionic Resin (Experimental): Bioactive Ionic Resin restoration is used to elevate the subgingival cervical margin in deep class II cavities before receiving cad/cam onlay restoration
  Interventions: Procedure: Bioactive Ionic Resin (cervical margin relocation)

INTERVENTIONS:
Procedure: Highly viscous glass ionomer (cervical margin relocation) — different dental restorative materials used to relocate deep cervical margins before receiving onlay restorations
  Arms: Highly viscous Glass Ionomer
Procedure: Low shrinkage Flowable Composite (cervical margin relocation) — different dental restorative materials used to relocate deep cervical margins before receiving onlay restorations
  Arms: Low shrinkage Flowable Composite
Procedure: Resin Modified Glass Ionomer (cervical margin relocation) — different dental restorative materials used to relocate deep cervical margins before receiving onlay restorations
  Arms: Resin Modified Glass Ionomer
Procedure: Bioactive Ionic Resin (cervical margin relocation) — different dental restorative materials used to relocate deep cervical margins before receiving onlay restorations
  Arms: Bioactive Ionic Resin

SUMMARY:
The current study intends to evaluate the effect of cervical margin relocation with different restorative materials on three-year clinical performance of indirect Computer-Aided-Design (CAD)/ Computer-Aided-Manufacture (CAM) onlay restorations. This study is designed to test the null hypothesis that the three-year clinical performance of onlay restorations is significantly affected by cervical margin relocation with different restorative materials.

ELIGIBILITY:
Inclusion Criteria:

* Good general health
* Good oral hygiene
* Patient aging 20-40 y
* Patients with proximal deep carious lesion
* International caries detection and assessment system (ICDAS) 4 or 5 that diagnosed clinically and radiographically.
* Normal response to a vitality test.

Exclusion Criteria:

* poor general health
* poor oral hygiene
* Teeth would need direct pulp capping
* Teeth act as abutment for fixed or removable prosthesis.
* patients with excessive parafunctional habits
* Patient potentially unable to be compliant to recall visits

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 64 (Actual)
Dates: Start 2021-08-24 (Actual); Primary Completion 2022-01-05 (Actual); Study Completion 2025-01 (Estimated)

PRIMARY OUTCOMES:
Gingiva | three year follow up
  Gingival Index Scale from 0 to 3 will be used for evaluation considering that score 0 represents normal gigiva while score 3 represents severely inflamed gingiva
Modified World Dental Federation (FDI) clinical Criteria | three year follow up
  1. Functional Properties of restorations:
     1. Fracture of material and retention
     2. Marginal adaptation
     3. Radiographic examination
  2. Biological Properties of restorations
     1. Postoperative (hyper-sensitivity and tooth vitality
     2. Recurrence of caries
     3. Tooth integrity (enamel cracks, tooth fractures)
     4. Periodontal Response
     5. Adjacent mucosa
  Descriptive scale from 1 to 5. Note: 1 is clinically excellent 5 is clinically poor.
  Scores(1-3) are considered sufficient The overall cumulative success rate of restorations will be evaluated

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of dentistry , Mansoura University, Al Mansurah, Dakahlia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided